CLINICAL TRIAL: NCT01971515
Title: A Phase I, First-in-Human, Dose Escalation Trial of MSC2363318A, a Dual p70S6K/Akt Inhibitor, in Subjects With Advanced Malignancies
Brief Title: First-in-Human Dose Escalation Trial in Subjects With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR100018-001
Record Dates: First submitted 2013-10-23; First posted 2013-10-29 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Solid Tumor
Keywords: MSC2363318A; Maximum tolerated dose; Dose limiting toxicities; Recommended phase 2 dose; M2698; Metastatic Breast Cancer; HER2+ Metastatic Breast Cancer; Hormone refractory ER/PR+ breast cancer; Tamoxifen; PAM Pathway Alteration(s); PAM Pathway; Targeted Therapy; P70S6K; AKT Inhibition; PI3K Pathway; HER2+ Trastuzumab Resistance
MeSH Terms: conditions — Breast Neoplasms | interventions — M2698; Trastuzumab; Tamoxifen

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MSC2363318A (Experimental)
  Interventions: Drug: MSC2363318A
- MSC2363318A plus Trastuzumab (Experimental)
  Interventions: Drug: MSC2363318A plus Trastuzumab
- MSC2363318A plus Tamoxifen (Experimental)
  Interventions: Drug: MSC2363318A plus Tamoxifen

INTERVENTIONS:
Drug: MSC2363318A — Part 1: MSC2363318A will be administered orally once daily for repeated 21-day cycles until intolerable toxicity or disease progression. Additional dose escalations will continue until Maximum Tolerated Dose (MTD) is reached, the food effect will be investigated in a separate group.
  Part 2 (Cohort 1): MSC2363318A will be administered orally once daily for repeated 21-day cycles until intolerable toxicity or disease progression in subjects with PAM pathway alterations.
  Dose reductions or treatment interruptions will be made at the discretion of the Investigator. If treatment interruption is required due to an acute or less severe but intolerable MSC2363318A-related event, at least a 1-week break is recommended. If, at retreatment, the dose reduction is not required, then the "continuous daily dosing regimen" may be replaced with an "intermittent dose regimen" of 2 weeks on, 1 week off (i.e. daily dosing from Day 1 to Day 15 followed by no dosing on Day 16 to Day 21 of the cycle).
  Other Names: M2698
  Arms: MSC2363318A
Drug: MSC2363318A plus Trastuzumab — Part 2 Cohort 2: MSC2363318A will be administered orally once daily for repeated 21-day cycles in combination with Trastuzumab.
  Dose reductions or treatment interruptions will be made at the discretion of the Investigator. If treatment interruption is required due to an acute or less severe but intolerable MSC2363318A-related event, at least a 1-week break is recommended. If, at retreatment, the dose reduction is not required, then the "continuous daily dosing regimen" may be replaced with an "intermittent dose regimen" of 2 weeks on, 1 week off (i.e. daily dosing from Day 1 to Day 15 followed by no dosing on Day 16 to Day 21 of the cycle).
  Trastuzumab is a recombinant IgGI kappa humanized monoclonal antibody administered weekly by intravenous infusion.
  Arms: MSC2363318A plus Trastuzumab
Drug: MSC2363318A plus Tamoxifen — Part 2 Cohort 3: MSC2363318A will be administered orally once daily for repeated 21-day cycles in combination with Tamoxifen.
  Dose reductions or treatment interruptions will be made at the discretion of the Investigator. If treatment interruption is required due to an acute or less severe but intolerable MSC2363318A-related event, at least a 1-week break is recommended. If, at retreatment, the dose reduction is not required, then the "continuous daily dosing regimen" may be replaced with an "intermittent dose regimen" of 2 weeks on, 1 week off (i.e. daily dosing from Day 1 to Day 15 followed by no dosing on Day 16 to Day 21 of the cycle).
  Tamoxifen is a nonsteroidal antiestrogen administered daily by oral administration.
  Arms: MSC2363318A plus Tamoxifen

SUMMARY:
This is a Phase 1, first-in-human, open-label, non-randomized, dose escalation, trial to explore the safety, tolerability, pharmacokinetic (PK), pharmacodynamic (PD) and clinical activity signals of MSC2363318A.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to (>=)18 years
* Confirmed diagnosis of advanced malignancies that may be controlled with p70S6K or Akt inhibition based on already identified molecular alteration known to affect the PAM pathway, such as:: such as: such as: phosphate and tensin homolog (PTEN), phosphoinositide 3-Kinase catalytic subunit alpha isoform (PIK3CA), protein kinase B 1 (Akt 1), Akt 3, mammalian target of rapamycin (mTOR), tumor sclerosis complex 1 (TSC1), tumor sclerosis complex 2 (TSC2), in subjects who have received at least all treatment options considered to be standard therapy, unless some available treatment are not acceptable to the subject. For the dose escalation portion of the trial, subjects must have received the standard therapy unless intolerant or contraindicated.

  * Part 2, Cohort 1: For subjects with only PAM pathway alterations, subjects must have only PAM alterations, excluding Akt2 activating mutations or amplifications, and no other genomic alterations.
  * Part 2, Cohort 2: Histologically confirmed local laboratory testing (immunohistochemistry 3+ staining and/or fluorescence in situ hybridization ratio >= 2.0) HER2+ metastatic breast cancer subjects who are resistant to trastuzumab-containing treatment and progressed on trastuzumab, pertuzumab, a taxane, and/or trastuzumab emtansine. There is no limit regarding the number of prior lines of therapy. Subjects may be enrolled regardless of whether or not their tumor harbors a PAM pathway alteration (documentation of PAM pathway alteration for this cohort is not required).
  * Part 2, Cohort 3: Histologically and/or cytologically confirmed diagnosis of breast cancer with hormone receptor-positive status (ER and/or PgR positive) and HER2-negative status with prior exposure to tamoxifen and/or an aromatase inhibitor and/or an aromatase inhibitor plus palbociclib. Prior treatment with tamoxifen in the neoadjuvant setting is allowed but must have been discontinued for at least 1 year prior to the first dose.
* Measurable disease using clinically appropriate criteria for the type of malignancy, RECIST version 1.1 for solid tumors and Cheson 2007 for lymphoma
* A tumor accessible for biopsies and consent to undergo tumor biopsies before and during MSC2363318A treatment. Subjects who do not have a tumor suitable for biopsy (such as, but not limited to, high procedural risk, inaccessible site for needle biopsy, etc.) but are otherwise eligible for this study may be considered for enrollment on a case-by-case basis after discussion with the Medical Monitor of the study
* Ability to read and understand the informed consent form and willingness and ability to give informed consent and demonstrate comprehension of the trial before undergoing any trial activities
* Negative blood pregnancy test at the screening visit for women of childbearing potential
* Willingness to avoid pregnancy and breast feeding beginning two weeks before the first MSC2363318A dose and ending three months after the last trial treatment. Male subjects with female partners of childbearing potential and female subjects of childbearing potential must use adequate contraception in the judgment of the Investigator, such as a two barrier method or a one barrier method with spermicide or intrauterine device during trial treatment dosing and for 3 months after the last dose of the study.

Exclusion Criteria:

* Eastern Cooperative Oncology Group Performance Status >=2
* Previous therapy with:

  * Chemotherapy, immunotherapy, biologic therapy, or any other anticancer therapy within 2 weeks (or five elimination half lives for noncytotoxics, whichever is shorter) of Day 1 of trial drug treatment (6 weeks for nitrosureas or mitomycin). Subjects on therapy with trastuzumab (trastuzumab cohort) may continue with trastuzumab during the screening phase of the study. Subjects on endocrine therapy may continue with antihormonal therapy until Day 1 of the study.
  * Any investigational agent within 3 weeks of Day 1 of trial drug treatment
  * Extensive prior radiotherapy on more than 30 percent of bone marrow reserves, or prior bone marrow/stem cell transplantation within 5 years from enrolment
  * Palliative radiation therapy within 2 weeks of Day 1 of trial drug treatment
* Known tumor EGFR, KRAS, and/or Akt2 mutations or amplification
* Ongoing toxicity due to a prior therapy, unless returned to baseline or Grade 1. Grade 2 toxicities (e.g., alopecia or peripheral neuropathy) that are not likely to increase the subject's safety risk while receiving trial treatment may be accepted after Sponsor approval.
* Major surgical intervention or participation in a therapeutic clinical trial within 28 days from Day 1 of the first dose of MSC2363318A
* Bone marrow impairment, renal impairment, liver function abnormality and impaired cardiac function as defined in the protocol
* History of cerebral vascular accident or stroke within the previous 2 years
* Uncontrolled hypertension
* History of Grade 3 or 4 allergic reactions attributed to compounds of similar chemical or biologic composition as MSC2363318A
* Known symptomatic central nervous system (CNS) metastases
* History of difficulty swallowing, malabsorption or other chronic gastrointestinal disease or conditions that may hamper compliance and/or absorption of the investigational product
* Known human immunodeficiency virus, viral hepatitis, or tuberculosis positivity
* Legal incapacity or limited legal capacity
* Any other condition which, in the opinion of the Investigator, might impair the subject's tolerance of trial treatment, the safety of the individual subject or the outcome of the trial. (including but not limited to: history of major depressive episode, bipolar disorder, obsessive-compulsive disorder, schizophrenia, suicidal attempt or ideation, homicidal ideation, or >= Common Terminology Criteria for Adverse Events [CTCAE] Grade 3 anxiety)
* Immediate prior therapy with a PAM pathway inhibitor (i.e., the subject is excluded if the last treatment regimen, prior to MSC2363318A, was a PAM pathway inhibitor, or if the last PAM pathway inhibitor that the subject was treated with occured less than 2 months prior to Day 1 of trial drug treatment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2013-12-13 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-09 (Actual)

PRIMARY OUTCOMES:
Number of dose limiting toxicities (DLTs) in Dose Escalation and Trastuzumab or Tamoxifen combination arms | Up to Day 21 of Cycle 1
Number of subjects with Treatment-emergent adverse events (TEAEs), Serious Adverse Events (SAEs), and deaths in cohort for subjects with PAM pathway alterations | Baseline up to Day 30 after the last dose of study treatment

SECONDARY OUTCOMES:
Observed Maximum Plasma Concentration (Cmax) | Days 1, 2, 8 and 15 of Cycle 1 and Days 1, 8 and 15 of Cycle 2, Cycle 3
Time To Reach Maximum Plasma Concentration (Tmax) | Days 1, 2, 8 and 15 of Cycle 1 and Days 1, 8 and 15 of Cycle 2, Cycle 3
Area Under Plasma Concentration Versus Time Curve From Time Zero to Last Sampling Time (AUC0-t) | Days 1, 2, 8 and 15 of Cycle 1 and Days 1, 8 and 15 of Cycle 2, Cycle 3
Area Under the Plasma Concentration Versus Time Curve From Time Zero to Infinity (AUC0-inf) | Days 1, 2, 8 and 15 of Cycle 1 and Days 1, 8 and 15 of Cycle 2, Cycle 3
Area Under Plasma Concentration Versus Time Curve Within One Dosing Interval (AUCtau) | Days 1, 2, 8 and 15 of Cycle 1 and Days 1, 8 and 15 of Cycle 2, Cycle 3
Apparent Terminal Half-life ( t1/2) | Days 1, 2, 8 and 15 of Cycle 1 and Days 1, 8 and 15 of Cycle 2, Cycle 3
Apparent Oral Clearance (CL/F) | Days 1, 2, 8 and 15 of Cycle 1 and Days 1, 8 and 15 of Cycle 2, Cycle 3
Apparent Oral Clearance Steady State (CLss/F) | Days 1, 2, 8 and 15 of Cycle 1 and Days 1, 8 and 15 of Cycle 2, Cycle 3
Apparent Volume of Distribution (Vz/F) | Days 1, 2, 8 and 15 of Cycle 1 and Days 1, 8 and 15 of Cycle 2, Cycle 3
Apparent Volume of Distribution at Steady State (Vss/F) | Days 1, 2, 8 and 15 of Cycle 1 and Days 1, 8 and 15 of Cycle 2, Cycle 3
Factor to Assess the Increase of Drug Concentration in Plasma Until Steady State is Reached [Racc(AUC)] | Days 1, 2, 8 and 15 of Cycle 1 and Days 1, 8 and 15 of Cycle 2, Cycle 3
Factor to Assess the Maximal Increase of Drug Concentration in Plasma [Racc (Cmax)] | Days 1, 2, 8 and 15 of Cycle 1 and Days 1, 8 and 15 of Cycle 2, Cycle 3
Number of subjects with best overall response according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v 1.1) or Cheson 2007 | Evaluation were performed on Day 1 of every alternate cycle until tumor progression
Percentage of subjects with clinical benefit | Week 12
  Percentage of subjects with clinical benefit is defined as subjects with complete response (CR) or partial response (PR) at week 12, based on tumor assessment as determined by RECIST version 1.1 or Cheson 2007.
Disease control rate (DCR) for Cohort 2 only | Week 6
Progression-free survival (PFS) rate for Cohorts 2 and 3 only | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono, Inc., Rockland MA, a subsidiary of Merck KGaA, Darmstadt, Germany
Locations (15):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California at San Diego, Moores Cancer Center, San Diego, California
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Metairie Oncology, Metairie, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai, New York, New York
  - Medical University of South Carolina, Charleston, South Carolina
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Fletcher Allen Health Care, Inc., Burlington, Vermont

REFERENCES:
- [Derived] Tsimberidou AM, Shaw JV, Juric D, Verschraegen C, Weise AM, Sarantopoulos J, Lopes G, Nemunaitis J, Mita M, Park H, Ellers-Lenz B, Tian H, Xiong W, Kaleta R, Kurzrock R. Phase 1 study of M2698, a p70S6K/AKT dual inhibitor, in patients with advanced cancer. J Hematol Oncol. 2021 Aug 18;14(1):127. doi: 10.1186/s13045-021-01132-z. PMID 34407844